CLINICAL TRIAL: NCT06480669
Title: Impact of Intermittent Fasting and Mediterranean Diet on the Physical Health of the Elderly: A Randomized Controlled Trial
Brief Title: Impact of Intermittent Fasting and Mediterranean Diet on the Physical Health of the Elderly
Acronym: FASTMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, María Isabel Iguacel Azorín, Associate Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI23/610
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Diabetes; Hypertension; Dyslipidemias; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding (TRF) (Experimental): 8 participants who followed a 12/12 Time Restricted Feeding (12 consecutive hours of fasting, from 20:30 to approximately 8:30 the following day).
  Interventions: Other: Time Restricted Feeding
- Mediterranean diet (Active Comparator): A control group consisting of 9 participants who followed a standard Mediterranean diet.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Time Restricted Feeding — 8 participants who practiced a 12/12 TRF (12 hours of fasting, from approximately 20:30 to 8:30 the following day).
  Other Names: TRF
  Arms: Time Restricted Feeding (TRF)
Other: Mediterranean Diet — A control group consisting of 9 participants who followed a standard Mediterranean diet.
  Arms: Mediterranean diet

SUMMARY:
The prevalence of chronic diseases is increasing globally. In recent years, intermittent fasting has emerged as an effective dietary pattern against some of the most common chronic diseases in the elderly, alongside the Mediterranean diet.

The objective was to determine whether a 12-hour daily intermittent fasting regimen combined with a Mediterranean diet can improve analytical and anthropometric values in the elderly.

A total of 17 individuals of both sexes, over 60 years old, autonomous, and with preserved cognitive capacity participated. They were randomly divided into two groups: 8 people in the intervention group performed intermittent fasting along with a Mediterranean diet, and 9 in the control group adopted only a Mediterranean diet. The intervention lasted 3 months, with measurements taken at the beginning and end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age.
* Belong to the Bombarda health centre.
* Preserved cognitive capacity.
* Autonomy for basic and instrumental activities of daily living.
* Ability to follow a TRF and/or adopt a Mediterranean dietary pattern.

Exclusion Criteria:

* Underweight (BMI <18.5).
* Serious or chronic uncontrolled disease.
* Specific treatment that could alter blood and/or anthropometric values.
* Poorly controlled type 1 or type 2 insulin-dependent diabetes mellitus.
* Present or past episode of eating disorder (ED).
* High alcohol consumption.

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Biochemical values (mg/dL) | 12 weeks
  Basal glucose, High-Density Lipoprotein, Low-Density Lipoprotein, total cholesterol, triglycerides, serum transferrin, urea, uric acid, creatinine.
Blood Pressure (mmHg) | 12 weeks
  Blood pressure (Systolic blood pressure, diastolic blood pressure)
Anthropometric values (kg) | 12 weeks
  Weight
Anthropometric values (cm) | 12 weeks
  Weight, waist circumference, hip circumference.
Anthropometric values (kg/m^2) | 12 weeks
  Body mass index.
Anthropometric index (numerical rating scale) | 12 weeks
  Atherogenic index of plasma, waist/hip ratio.
Biochemical values (IU/L) | 12 weeks
  Alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase
Biochemical values (mg/L) | 12 weeks
  C-Reactive Protein
Biochemical values (µg/L) | 12 weeks
  Serum ferritin
Biochemical values (µg/dL) | 12 weeks
  Iron
Biochemical values (g/dL) | 12 weeks
  Albumin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No